CLINICAL TRIAL: NCT01864941
Title: Phase I/II Interventional Clinical Trial of Balloon Venoplasty for Chronic Cerebrospinal Venous Insufficiency in Multiple Sclerosis Patients
Brief Title: Interventional Clinical Trial for CCSVI in Multiple Sclerosis Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Multiple Sclerosis Society of Canada (Other)
Responsible Party: Principal Investigator, Anthony Traboulsee, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: H12-01153
Record Dates: First submitted 2013-05-13; First posted 2013-05-30 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; MS; CCSVI; Zamboni; catheter venography; balloon angioplasty
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Catheter Venography & Balloon Venoplasty (Active Comparator): Patients will undergo catheter venography with balloon venoplasty procedure.
  Interventions: Procedure: Catheter venography with balloon venoplasty; Device: Catheter venography with balloon venoplasty and balloon
- Catheter Venography Only (Sham Comparator): Patients will undergo catheter venography only.
  Interventions: Procedure: Catheter venography with balloon venoplasty

INTERVENTIONS:
Procedure: Catheter venography with balloon venoplasty — All eligible patients will undergo catheter venography with balloon venoplasty and/or sham at baseline and at week 48 (i.e. Cross over design) followed by clinical and radiologic observation for a minimum of 48 weeks after each procedure.
Device: Catheter venography with balloon venoplasty and balloon
  Arms: Catheter Venography & Balloon Venoplasty

SUMMARY:
To investigate the safety and tolerability of balloon venoplasty compared to sham in Multiple Sclerosis patients with Chronic Cerebrospinal Venous Insufficiency (CCSVI) as measured by adverse events occurring within 48 weeks of the procedure.

DETAILED DESCRIPTION:
Overview of study objectives are:

* To determine the safety and tolerability of venoplasty of CCSVI in Multiple Sclerosis (MS).
* To determine the short term and long term impact on validated patient measures and by physician and radiologic reported MS outcomes.
* To determine the short term and long term recurrence rate of CCSVI for veins that have been treated with venoplasty

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Relapsing Remitting Multiple Sclerosis (RRMS) or Secondary Progressive MS according to the McDonald criteria 2010
* Age 18 to 65 years inclusive
* Neurostatus (EDSS) score at screening from 0 to 6.5
* Fulfill ultrasound criteria for CCSVI

Exclusion Criteria:

* Previous venoplasty and/or stenting of extra cranial venous system

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2013-05; Primary Completion 2017-08-01 (Actual); Study Completion 2017-08-01 (Actual)

PRIMARY OUTCOMES:
Adverse Events | 48 weeks
  To investigate the safety and tolerability of balloon venoplasty compared to sham in Multiple Sclerosis (MS) patients with CCSVI as measured by adverse events occurring within 48 weeks of the procedure.

SECONDARY OUTCOMES:
Clinical Outcome | 48 weeks
  To evaluate the efficacy of balloon venoplasty compared to sham as reflected by patient reported quality of life, pain and fatigue scales 48 weeks after the procedure.
Clinical Outcome | 48 weeks
  To evaluate the efficacy of balloon venoplasty compared to sham as reflected by physician reported clinical scales 48 weeks after the procedure.
Clinical Outcome | 48 weeks
  To evaluate the efficacy of balloon venoplasty compared to sham as reflected by MRI 48 weeks after the procedure.
Clinical Outcome | 48 weeks
  To evaluate the efficacy of balloon venoplasty compared to sham as reflected by catheter venography 48 weeks after the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Traboulsee, MD, Study Director — University of British Columbia
Locations (4):
- Canada (4):
  - Vancouver Coastal Health - University of British Columbia Hospital, Vancouver, British Columbia
  - University of Manitoba Health Sciences Centre, Winnipeg, Manitoba
  - Centre Hospitalier de l'Université de Montréal, Montreal, Quebec
  - CHU de Québec - Hôpital de l'Enfant-Jésus, Québec, Quebec

REFERENCES:
- [Derived] Traboulsee AL, Machan L, Girard JM, Raymond J, Vosoughi R, Hardy BW, Emond F, Gariepy JL, Bone JN, Siskin G, Klass D, Isserow S, Illes J, Sadovnick AD, Li DK. Safety and efficacy of venoplasty in MS: A randomized, double-blind, sham-controlled phase II trial. Neurology. 2018 Oct 30;91(18):e1660-e1668. doi: 10.1212/WNL.0000000000006423. Epub 2018 Sep 28. PMID 30266886